CLINICAL TRIAL: NCT02876809
Title: A Model for Healthy Aging: Moscow Centenarians (AGE-100)
Acronym: AGE-100
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MCA-100
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Aging
Keywords: centenarians; geriatric; telomere length; progerin; metagenome; metabolome
MeSH Terms: conditions — Autosomal Emery-Dreifuss Muscular Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples with DNA will be taken for telomere lenth, metabolome and metagenome definition
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the associations between biomarkers of ageing, comprehensive geriatric status, telomere length and progerin level, the composition of the gut microbiota, 16sRNA metagenome sequencing in Moscow centenarians.

DETAILED DESCRIPTION:
The global average life expectancy and the average age of the population are growing steadily along with the age-related diseases. The same trend is also observed in our country. Although, maximum life span in Russia decreases. E.g., the number of centenarians in Moscow decreased by 244 persons from 2013 to 2014. There were about 400 centenarians in Moscow in 2014. That is about 3.3 per 100 000 population. In the US, this figure is about 10-20, and there are 50 centenarians per 100 000 population in the Okinawa region, Japan. The rate of ageing varies substantially, a prime example of this is the centenarians population. These people break conventional stereotypes about aging. Chronic diseases in centenarians are postponed. They are more active, they work longer, they can better tolerate stressful situations. Scientists all over the world are trying to find the secret of their longevity. Studies on the medical and social aspects of centenarian longevity are actively carried out in the US, Europe, Japan, Australia. In Russia studies were carried out in St. Petersburg, Western and Eastern Siberia. According to the New England Centenarian Study, the supercentenarians (persons who have lived more than 110 years) life span is actually equal to the healthy span without serious illnesses. The aim of research is to study features of social status, lifestyle, habits, clinical status, blood chemistry, the amount of progerin, genome, composition of the gut microbiota in Moscow centenarians in order to create a model of healthy aging. In this study a comprehensive analysis of the longevity phenomenon of one hundred centenarians from Moscow and the Moscow region planning to be conducted. Analyzing of anamnesis vitae, medical, social, neuro-cognitive, and genetic features is planning. Each study participant will undergo a comprehensive geriatric assessment, including examination by the neurologist, an assessment of cognitive status,psychogeriatric consultation with the assessment of self-perceptions of aging and depression assessment by using the geriatric depression scale, neuropsychological testing using the Montreal Cognitive Assessment (MoCA), verbal recognition memory 12 word test, clock-drawing test.Telomere length and progerin level in buffy coat layer evaluation, 16sRNA metagenome sequencing, and nuclear magnetic resonance spectroscopy for qualitative and quantitative analysis of metabolites in blood serum, will be done in all participants. This study will take the science closer to the goal of identifying the patterns of "healthy" aging.

ELIGIBILITY:
Inclusion Criteria:

age over 90 years

-

Exclusion Criteria:

age under 90 years refusal to participate in the study

-

Min Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population consists of 100-age Moscow long-livers chosen according to data of Moscow clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Definition of frailty prevalence among 100-Centenarians | 0 month
  Frailty will be measured by comprehensive geriatric assessment, including examination by the neurologist, an assessment of cognitive status,psychogeriatric consultation with the assessment of self-perceptions of aging and depression assessment by using the geriatric depression scale, neuropsychological testing using the Montreal Cognitive Assessment (MoCA), verbal recognition memory 12 word test, clock-drawing test

SECONDARY OUTCOMES:
Definition of telomere biology status | 0 month
  Relative telomere length in genomic DNA and telomerase activity in monocytes will be assessed by real-time PCR.
Definition of vascular aging | 0 month
  Vascular aging will be measured by intima-media thickness measurement and plaque presence determination by ultrasonography in both left and right common carotid arteries. Arterial stiffness will be assess by aortic pulse wave velocity measuring by SphygmoCor.

CONTACTS AND LOCATIONS:
Overall Officials: Olga N. Tkacheva, Professor, Principal Investigator — Russian Gerontology Clinical Research Center
Locations (1):
- Pirogov Russian National Research Medical University of the Ministry of Health of the Russian Federation, Russian Gerontology Clinical Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This novel approach support the hypothesis that a complex remodeling of lipid, amino acid metabolism, and of gut microbiota functionality are key regulatory processes marking exceptional longevity in humans. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Collino+S%2C+Montoliu+I%2C+Martin+FP%2C+Scherer+M%2C+Mari+D%2C+Salvioli+S%2C+et+al.+Metabolic+signatures+of+extreme+longevity+in+northern+Italian+centenarians+reveal+a+complex+remodeling+of+lipids%2C+amino+acids%2C+and+gut+microbiota+metabolism.
- See also: While some centenarians have poor health and functioning upon reaching age 100, others are able to achieve exceptional longevity in relatively good health and without loss of functioning. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Ailshire+JA%2C+Beltran-Sanchez+H%2C+Crimmins+EM.+Becoming+centenarians%3A+disease+and+functioning+trajectories+of+older+US+Adults+as+they+survive+to+100.+J+Gerontol+A+Biol+Sci+Med+Sci
- See also: Available data indicate improved DNA repair and antioxidant defense mechanisms in "super old" humans, which are comparable with much younger cohorts. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Franzke+B%2C+Neubauer+O%2C+Wagner+KH.+Super+DNAging-New+insights+into+DNA+integrity%2C+genome+stability+and+telomeres+in+the+oldest+old.+Mutat+Res+Rev+Mutat+Res
- See also: Results suggest that a better preservation of DNA methylation status, a slower cell growing/metabolism, and a better control in signal transmission through epigenetic mechanisms may be involved in the process of human longevity. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Gentilini+D%2C+Mari+D%2C+Castaldi+D%2C+Remondini+D%2C+Ogliari+G%2C+Ostan+R%2C+et+al.+Role+of+epigenetics+in+human+aging+and+longevity%3A+genome-wide+DNA+methylation+profile+in+centenarians+and+centenarians%27+offspring